CLINICAL TRIAL: NCT01741324
Title: Comparing Different Amounts of Vitamin D Supplementation to Preschool Children Living in Northern and Southern Sweden
Acronym: Dvisum
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Umeå University (Other)
Collaborators: Region Skane (Other)
Responsible Party: Principal Investigator, Torbjörn Lind, Associate professor, Umeå University
Allocation: Randomized | Model: Factorial | Masking: Quadruple | Purpose: Prevention
Other Study IDs: Dvisum
Record Dates: First submitted 2012-11-26; First posted 2012-12-04 (Estimated); Last update posted 2016-11-01 (Estimated); Status verified 2016-10

CONDITIONS: Vitamin D Deficiency
MeSH Terms: conditions — Vitamin D Deficiency

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (10):
- Umeå, vitamin D 25 microg/d, light skin (Experimental): Participants with light skin will be randomized to a milk drink providing 25 microg vitamin D3 per day.
  Interventions: Dietary Supplement: Vitamin D 25 microg/d
- Umeå, vitamin D 10 microg/d, dark skin (Active Comparator): Participants with dark skin will be randomized to a milk drink providing 10 microg vitamin D3 per dag.
  Interventions: Dietary Supplement: Vitamin D 10 microg/d
- Umeå, vitamin D 10 microg/d, light skin (Active Comparator): Participants with light skin will be randomized to a milk drink providing 10 microg vitamin D3 per dag.
  Interventions: Dietary Supplement: Vitamin D 10 microg/d
- Malmö, vitamin D 25 microg/d, dark skin (Experimental): Participants with dark skin will be randomized to a milk drink providing 25 microg vitamin D3 per day.
  Interventions: Dietary Supplement: Vitamin D 25 microg/d
- Malmö, vitamin D 25 microg/d, light skin (Experimental): Participants with light skin will be randomized to a milk drink providing 10 microg vitamin D3 per day.
  Interventions: Dietary Supplement: Vitamin D 25 microg/d
- Malmö, vitamin D 10 microg/d, dark skin (Active Comparator): Participants with dark skin will be randomized to a milk drink providing 10 microg vitamin D3 per day.
  Interventions: Dietary Supplement: Vitamin D 10 microg/d
- Malmö, vitamin D 10 microg/d, light skin (Active Comparator): Participants with light skin will be randomized to a milk drink providing 10 microg vitamin D3 per day.
  Interventions: Dietary Supplement: Vitamin D 10 microg/d
- Malmö, placebo, dark skin, (Placebo Comparator): Participants with dark skin will be randomized to a milk drink without added vitamin D (placebo).
  Interventions: Dietary Supplement: No extra vitamin D
- Malmö, placebo, light skin (Placebo Comparator): Participants with light skin will be randomized to a milk drink without added vitamin D (placebo).
  Interventions: Dietary Supplement: No extra vitamin D
- Umeå, vitamin D 25 microg/d, dark skin (Experimental): Participants with dark skin will be randomized to a milk drink providing 25 microg vitamin D3 per day.
  Interventions: Dietary Supplement: Vitamin D 25 microg/d

INTERVENTIONS:
Dietary Supplement: Vitamin D 25 microg/d — The vitamin D supplement will be provided as a milk drink taken daily.
  Arms: Malmö, vitamin D 25 microg/d, dark skin; Malmö, vitamin D 25 microg/d, light skin; Umeå, vitamin D 25 microg/d, dark skin; Umeå, vitamin D 25 microg/d, light skin
Dietary Supplement: Vitamin D 10 microg/d — The vitamin D supplement will be provided as a milk drink taken daily.
  Arms: Malmö, vitamin D 10 microg/d, dark skin; Malmö, vitamin D 10 microg/d, light skin; Umeå, vitamin D 10 microg/d, dark skin; Umeå, vitamin D 10 microg/d, light skin
Dietary Supplement: No extra vitamin D — Milk drink with no extra vitamin D (placebo)
  Other Names: Placebo
  Arms: Malmö, placebo, dark skin,; Malmö, placebo, light skin

SUMMARY:
Vitamin D has a range of biological effects of public health relevance. Vitamin D status is assessed on levels of its metabolite 25-hydroxyvitamin D [25(OH)D], where levels < 50 nmol/L indicate insufficiency. Despite studies indicating that the vitamin D intake among Swedish children are significantly below recommendations, little is known of their vitamin D status. The investigators have recently found inadequate vitamin D status in pre-school children living in northern Sweden, especially in dark-skinned children and during the winter months despite vitamin D intakes meeting the recommendations. Overall, 25% of the light skinned and 40% of the dark skinned children had S-25(OH) D <50 nmol/L (Öhlund I, unpublished data). The aim is to examine which amount of vitamin D is needed to maintain or increase S-25(OH)D to ≥50 nmol/L among 97.5% of the participants regardless of skin color or geographic location (northern or southern Sweden). Furthermore the investigators will examine if vitamin D status affects on health markers as bone density, blood pressure, serum lipids, fatty acids, inflammatory and immunological markers and mental wellbeing.

Children aged 5-8 years living either northern (Umeå) or southern Sweden (Malmö) will be recruited to this trial during November-December 2012. They will be randomized to a vitamin D supplement of either 10 or 25 g per day, or in Malmö also placebo to be used for three months. The randomization will be stratified according to skin color (light or dark) according to a method using visual inspection and interviews of parents/guardians. The investigators will use a 2×2×2 factorial design to investigate the effects of two different doses of vitamin D (10 µg and 25 µg) in children with dark and light skin color, living in northern (Umeå) and southern (Malmö), Sweden. In order to achieve a moderate difference between groups (effect size 0.25) 20 children per group are required (power> 87%, alpha = 0.05). With an estimated dropout of 10%, a total of 220 children will be included.

At baseline, the participants will undergo blood sampling for S-25(OH)D and other biomarkers, blood pressure and anthropometrical measurements, including bone densitometry and body composition using air displacement pletysmography, and the parents will answer a questionnaire on behavioral and emotional problems in the participating child using the Child Behavior Checklist. These measurements will be repeated at follow-up in February-March 2013.

DETAILED DESCRIPTION:
Vitamin D has a range of biological effects of public health relevance (Prentice et al, 2008). Besides its well known role in mineralization of bone and teeth, vitamin D also play important roles in metabolic functions, the pathogenesis of certain diseases, e.g. type 1 diabetes, celiac disease, asthma and allergies, as well as in the prevention of cancer (Holick, 2008).

Vitamin D status is assessed on plasma or serum levels of its metabolite 25-hydroxyvitamin D [25(OH)D, calcidiol] as it reflects the sum of vitamin D converted in the skin through sunlight exposure and from dietary sources. Several reports advocate that levels <37 nmol/L denote severe vitamin D deficiency; levels <50 nmol/L insufficient; 50-75 nmol/L suboptimal levels and ≥75nmol/L optimal levels (Dawson-Hughes et al, 2005, Huh et al, 2008, Yetley, 2008). In children, most suggested cut-off values for adequate levels of 25(OH)D are based on the absence of rickets, increased measures of bone mineralization and maximal suppression of parathyroid hormone (PTH) levels (Greer, 2009).

The major source of vitamin D is dermal biosynthesis catalyzed by ultraviolet B sunlight (Cashman et al, 2011). However, during winter, northern Sweden has limited hours of daylight leading to reduced sun exposure. Consequently, the dietary source of vitamin D is of specific importance in this region (Brustad et al, 2007, Edvardsen et al, 2007). Fatty fish, eggs, vitamin D fortified milk and margarines are the main sources, mainly supplying the most active form D3. These are important basic foods which also contain common food allergens. Thus, children with food allergies to milk, fish, and egg can be at increased risk of vitamin D deficiency. Several dairy products are fortified with vitamin D, but in some products in the form of D2 which is not as bioactive as D3.

Skin color affects the capacity to form vitamin D3 as children with dark complexion need 5-10 times more sun exposure to generate the same amount of vitamin D3 compared to fair-skinned children, and therefore are at increased risk of vitamin D deficiency when exposure to sun is limited (Holick, 2005). Recently the recommendations on protecting the skin from sunshine to reduce the risk of skin cancer later in life has been debated as it may increase the risk of vitamin D deficiency (Stechschulte et al, 2011). Obesity in children might be another risk factor for vitamin D deficiency, since an increased proportion of available vitamin D may be stored in adipose tissue thus lowering the S-25(OH)D (Prentice, 2008).

Despite studies indicating that the vitamin D intake among Swedish children and adolescents are significantly below recommendations, little is known of their vitamin D status (Garemo et al, 2007, Enghardt et al, 2006, Öhlund et al, 2010). Furthermore there is a paucity of studies investigating vitamin D intake and status in food-allergic adolescents who may be at increased risk of vitamin D insufficiency due to strict avoidance of vitamin D containing foods.

Recently the investigators of Dvisum assessed Vitamin D status in pre-school children (n=90; mean age 54+/-7.1 mo), all living in northern Sweden (latitude 63°) and half of them with fair skin, half with darker complexion. The study group was examined first in August-September (late summer) and then the following January-February (winter). Skin type, vitamin D intake, anthropometrics, S-25(OH) D and parathyroid hormone (S-PTH) were assessed. The investigators found inadequate vitamin D status in these children living in northern Sweden, especially in dark-skinned children and during the winter despite vitamin D intakes meeting the recommendations, prompting strategies to improve intake of vitamin D in this population. Overall, 25% and 40% of the light and dark skinned had S-25(OH) D <50 nmol/L.

The aim is to examine which amount of vitamin D is needed to maintain or increase S-25(OH)D to ≥50 nmol/L among 97.5% of the participants regardless of skin color or geographic location (northern or southern Sweden). Furthermore the investigators will examine if vitamin D status affects health markers such as bone density, blood pressure, serum lipids, fatty acids and inflammatory and immunological markers and mental wellbeing.

In order to identify whether there are differences depending on the latitude within Sweden, children will be recruited both from northern Sweden (Umeå) and from southern Sweden (Malmo). As it is unclear what levels of the serological marker 25 (OH) D that affect the health of children, different markers of health will be examined before and after the intervention. Children aged 5-8 years, 50% fair-skin 50 % darker skin, in northern Sweden (Umeå) and southern Sweden (Malmö) will be included in a longitudinal, randomized trial. The children are first examined in November-December and randomized to a vitamin D supplement of either 10 or 25 g per day, to be used for three months. At the follow up in February-March all examinations will be repeated.

The investigators will use a 2 × 2 × 2 factorial design to investigate the effects of two different doses of vitamin D (10 µg and 25 µg) in children with dark and light skin color, living in northern (Umeå) and southern (Malmö), Sweden. In order to achieve a moderate difference between groups (effect size 0.25) requires 20 children per group (power>87%, alpha = 0.05). With this group size, we can see a group difference in the S-25 (OH) D of 3.75 nmol/L, S-PTH of 0.35 mmol/L and bone mineral density in the lumbar region of 0.075 g/cm2. In Skåne, but not Umeå also a placebo group will participate. With an estimated dropout of 10%, a total of 220 children will be included.

The study include sampling for analysis of S-25 (OH) D, calcium, phosphate, alkaline phosphatase (ALP), magnesium, PTH and osteocalcin, serum lipids (total cholesterol, HDL cholesterol, LDL cholesterol. ApoA1 and ApoB lipoprotein) and fatty acids as well as inflammatory and immunological markers (CRP, interleukin (IL) -1 and 2, IL-4, IL-6, I-10, Il-17, CD40 ligand, TNF and IFNγ, fibrinogen and antisecretory factor). Before sampling, the children receive a topical anesthetic (EMLA).

Measurements of blood pressure and anthropometric measurements of length, weight, waist circumference and bone densitometry (DEXA) and body composition (fat mass% and fat free mass) using a Air Displacement Plethysmography ( BOD POD) Questions about diet, vitamin supplements, foreign travel, how much time the children spend time outdoors and the use of sunscreen as well as questions about the child's health and family situation will be answered by the parents through a questionnaire. To investigate the possible association between vitamin D status and mental well-being, the investigators will use the Child Behaviour Checklist (CBCL).

This study is national with a multicultural perspective, it is expected to provide knowledge about the needs of vitamin D to prevent vitamin D deficiency. The study is also expected to provide a better understanding of association between vitamin D status and various markers of health among children.

By preventing vitamin D deficiency, poor bone development, susceptibility to infections, and perhaps prone to autoimmune diseases and cardiovascular risk factors could be reduced, and hopefully the mental well-being improved, which reduces costs to both society and the individual, and reduces unnecessary suffering of individuals.

ELIGIBILITY:
Inclusion Criteria:

* 5-7 years of age
* Healthy

Exclusion Criteria:

* Chronic illness, including coeliac disease or other chronic gastrointestinal disorders
* Drugs that can affect bone health or vitamin D uptake
* Cow's milk allergy

Ages: 5 Years to 7 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 220 (Actual)
Dates: Start 2012-11; Primary Completion 2013-04 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Serum 25OH-vitamin D levels | 90 days after start of treatment

SECONDARY OUTCOMES:
Bone mineralisation | 120 days after start of treatment
  Bone mineralisation will be measured with DXA-scan, serum PTH and serum osteocalcin

OTHER OUTCOMES:
Inflammatory and immunological markers | 90 days after start of treatment
  CRP, interleukin (IL) -1 and 2, IL-4, IL-6, I-10, Il-17, CD40 ligand, TNF-alfa, IFNγ, fibrinogen and antisecretory factor
Behavioral and emotional well-being | 90 days after start of treatment
  Parental assessment using Child Behavioral Checklist

CONTACTS AND LOCATIONS:
Overall Officials: Inger Öhlund, Ph.D., Principal Investigator — Umeå University; Torbjörn Lind, M.D., Ph.D., Study Chair — Umeå University; Pia Karlsland-Åkesson, M.D., Ph.D., Study Chair — University hospital, Malmö/Lund; Sven-Arne Silfverdal, M.D., Ph.D., Study Chair — Umeå University; Olle Hernell, M.D., Ph.D., Study Chair — Umeå University
Locations (2):
- Sweden (2):
  - Department of Pediatrics, University hospital Malmö, Malmo, Skåne County
  - Pediatrics, Department of Clinical Sciences, Umeå University, Umeå, Västerbotten County

REFERENCES:
- [Background] Prentice A, Goldberg GR, Schoenmakers I. Vitamin D across the lifecycle: physiology and biomarkers. Am J Clin Nutr. 2008 Aug;88(2):500S-506S. doi: 10.1093/ajcn/88.2.500S. PMID 18689390
- [Background] Holick MF. The vitamin D deficiency pandemic and consequences for nonskeletal health: mechanisms of action. Mol Aspects Med. 2008 Dec;29(6):361-8. doi: 10.1016/j.mam.2008.08.008. Epub 2008 Sep 2. PMID 18801384
- [Background] Dawson-Hughes B, Heaney RP, Holick MF, Lips P, Meunier PJ, Vieth R. Estimates of optimal vitamin D status. Osteoporos Int. 2005 Jul;16(7):713-6. doi: 10.1007/s00198-005-1867-7. Epub 2005 Mar 18. PMID 15776217
- [Background] Huh SY, Gordon CM. Vitamin D deficiency in children and adolescents: epidemiology, impact and treatment. Rev Endocr Metab Disord. 2008 Jun;9(2):161-70. doi: 10.1007/s11154-007-9072-y. Epub 2008 Jan 4. PMID 18175220
- [Background] Yetley EA. Assessing the vitamin D status of the US population. Am J Clin Nutr. 2008 Aug;88(2):558S-564S. doi: 10.1093/ajcn/88.2.558S. PMID 18689402
- [Background] Greer FR. Defining vitamin D deficiency in children: beyond 25-OH vitamin D serum concentrations. Pediatrics. 2009 Nov;124(5):1471-3. doi: 10.1542/peds.2009-2307. Epub 2009 Oct 26. No abstract available. PMID 19858159
- [Background] Cashman KD, FitzGerald AP, Viljakainen HT, Jakobsen J, Michaelsen KF, Lamberg-Allardt C, Molgaard C. Estimation of the dietary requirement for vitamin D in healthy adolescent white girls. Am J Clin Nutr. 2011 Mar;93(3):549-55. doi: 10.3945/ajcn.110.006577. Epub 2011 Jan 26. PMID 21270380
- [Background] Brustad M, Edvardsen K, Wilsgaard T, Engelsen O, Aksnes L, Lund E. Seasonality of UV-radiation and vitamin D status at 69 degrees north. Photochem Photobiol Sci. 2007 Aug;6(8):903-8. doi: 10.1039/b702947k. Epub 2007 Jun 27. PMID 17668121
- [Background] Edvardsen K, Brustad M, Engelsen O, Aksnes L. The solar UV radiation level needed for cutaneous production of vitamin D3 in the face. A study conducted among subjects living at a high latitude (68 degrees N). Photochem Photobiol Sci. 2007 Jan;6(1):57-62. doi: 10.1039/b613263d. Epub 2006 Nov 10. PMID 17200737
- [Background] Holick MF. The vitamin D epidemic and its health consequences. J Nutr. 2005 Nov;135(11):2739S-48S. doi: 10.1093/jn/135.11.2739S. PMID 16251641
- [Background] Stechschulte SA, Kirsner RS, Federman DG. Sunscreens for non-dermatologists: what you should know when counseling patients. Postgrad Med. 2011 Jul;123(4):160-7. doi: 10.3810/pgm.2011.07.2315. PMID 21681000
- [Background] Prentice A. Vitamin D deficiency: a global perspective. Nutr Rev. 2008 Oct;66(10 Suppl 2):S153-64. doi: 10.1111/j.1753-4887.2008.00100.x. PMID 18844843
- [Background] Garemo M, Lenner RA, Strandvik B. Swedish pre-school children eat too much junk food and sucrose. Acta Paediatr. 2007 Feb;96(2):266-72. doi: 10.1111/j.1651-2227.2007.00093.x. PMID 17429918
- [Background] Enghardt B, Pearson M, Becker W. Dietary habits and nutrient intake in Swedish children 4 years old and school children in grade 2 and 5 (Riksmaten - barn 2003). Uppsala: National Food Administration (Livsmedelsverket), Uppsala, Sweden; 2006.
- [Background] Ohlund K, Olsson C, Hernell O, Ohlund I. Dietary shortcomings in children on a gluten-free diet. J Hum Nutr Diet. 2010 Jun;23(3):294-300. doi: 10.1111/j.1365-277X.2010.01060.x. Epub 2010 Mar 23. PMID 20337845
- [Derived] Ohlund I, Lind T, Hernell O, Silfverdal SA, Liv P, Karlsland Akeson P. Vitamin D status and cardiometabolic risk markers in young Swedish children: a double-blind randomized clinical trial comparing different doses of vitamin D supplements. Am J Clin Nutr. 2020 Apr 1;111(4):779-786. doi: 10.1093/ajcn/nqaa031. PMID 32140704
- [Derived] Karlsland Akeson P, Akesson KE, Lind T, Hernell O, Silfverdal SA, Ohlund I. Vitamin D Intervention and Bone: A Randomized Clinical Trial in Fair- and Dark-skinned Children at Northern Latitudes. J Pediatr Gastroenterol Nutr. 2018 Sep;67(3):388-394. doi: 10.1097/MPG.0000000000002031. PMID 29851760
- [Derived] Gyll J, Ridell K, Ohlund I, Karlsland Akeson P, Johansson I, Lif Holgerson P. Vitamin D status and dental caries in healthy Swedish children. Nutr J. 2018 Jan 16;17(1):11. doi: 10.1186/s12937-018-0318-1. PMID 29338758
- [Derived] Ohlund I, Lind T, Hernell O, Silfverdal SA, Karlsland Akeson P. Increased vitamin D intake differentiated according to skin color is needed to meet requirements in young Swedish children during winter: a double-blind randomized clinical trial. Am J Clin Nutr. 2017 Jul;106(1):105-112. doi: 10.3945/ajcn.116.147108. Epub 2017 Jun 14. PMID 28615261